CLINICAL TRIAL: NCT05575310
Title: Central Sesitization in Patients with Persistent Postsurgical Pain After a Knee Arthroplasty: a Prospective, Case Control, Observational Study
Brief Title: Central Sensitization in Total Knee Arthroplasty Patients with Persistent Pain
Status: Completed | Type: Observational
Sponsor: University of Barcelona (Other)
Collaborators: Consorci Hospitalari de Vic (Other); University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Marc Terradas Monllor, Dr. Marc Terradas-Monllor, University of Barcelona
Other Study IDs: CS-TKA
Record Dates: First submitted 2022-09-17; First posted 2022-10-12 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Pain, Chronic Postsurgical; Knee Osteoarthritis; Sensitization, Central
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- No Persistent Post Surgical Pain: The grouping variable will be the presence or not of persistent post-surgical pain. This will be a dichotomous variable obtained from the evaluation of pain intensity at 3 months after surgery. The tool used will be a 100mm Visual Analog Scale (VAS) (0 = no pain, 100 = worst pain imaginable) (25). Those with a VAS < 30 will be considered as patients with no persistent pain, while those with a VAS ≥ 30 will be considered as patients with persistent pain. This cut-off point has been determined by numerous authors in previous studies.
  Interventions: Procedure: Total Knee Arthroplasty
- Persistent Post Surgical Pain: While those with a VAS ≥ 30 will be considered as patients with persistent pain. This cut-off point has been determined by numerous authors in previous studies
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Articular knee surface replacement

SUMMARY:
Persistent post-surgical pain is a significant adverse effect after total knee arthroplasty, present in around 20% of the patients. Central sensitization may contribute to developing and maintaining pain. Therefore studies should investigate if pain processing altered mechanisms are present in this population.

DETAILED DESCRIPTION:
Numerous studies suggest that peripheral and central sensitization in patients with symptomatic knee osteoarthritis could be an important factor capable of explaining part of these poor outcomes after knee arthroplasty. Quantitative sensory testing has been frequently used to investigate this sensitization of the central nervous system and assess pain hypersensitivity locally and away from the affected region in patients with chronic knee osteoarthritis pain. Pressure algometry is a method described to determine pain thresholds to pressure and thus evaluate the sensitivity to pain due to tissue pressure. However, another aspect associated with sensitization is the downward modulation of peripheral inputs. This occurs in neurons in the posterior horn of the medulla and can be either inhibitory or facilitatory. The conditioned pain modulation test is a manifestation of this phenomenon, which can be easily assessed in patients, and is characterized by the modification of the response to the application of a painful stimulus when a second conditioning painful stimulus is applied. Conditioned pain modulation has been shown to be altered in patients with symptomatic knee osteoarthritis.

The literature suggests that although one of the main components of pain perpetuation with people with knee osteoarthritis is sensitization of the nervous system, successful knee arthroplasty is able to normalize its functioning. This implies that the maintenance of sensitization can be triggered by peripheral nociceptive stimuli. When performing a knee arthroplasty, the structures capable of generating these peripheral nociceptive stimuli are eliminated, so that the pain-generating mechanisms cannot be the same as before in those who manifest persistent post-surgical pain. For this reason, one of the hypotheses is that the mechanism responsible for causing this pain is a central mechanism and not a peripheral one. Although this hypothesis has not been fully tested, there are indications that people with chronic post-surgical pain may suffer peripheral and central sensitization processes, very similar to those that can be observed in people with symptomatic osteoarthritis of the knee that is not operated on, even though the structures involved are no longer present. This fact reinforces the theory of the involvement of a central mechanism in the perpetuation of pain after surgery.

Therefore, the present study aims to investigate the involvement of the central sensitization process in the perpetuation of postoperative pain in individuals undergoing total knee arthroplasty for primary symptomatic knee osteoarthritis. From a clinical point of view, current postoperative treatments focus mainly on improving the patient's functional outcomes (e.g., physical function and joint range of motion), and the status of the descending pain modulator system is rarely taken into account. The present study seeks to place importance on the central mechanisms in the perpetuation of pain after knee arthroplasty, to inspire new treatment protocols that take these processes into account.

ELIGIBILITY:
Inclusion criteria:

- Patients who underwent total knee arthroplasty due to painful primary osteoarthritis.

Exclusion criteria:

* Patients operated due to a revision surgery.
* Patients with a unicompartmental knee arthroplasty
* Pateints operated due to a fracture.
* Patients planning to undergo another lower extremity operation during the following 12 months.
* Patients with inflammatory or rheumatic diseases such as: rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus or ankylosing spondylitis.
* Patients with mental health conditions and/or major depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent total knee arthroplasty due to symptomatic, end-stage knee ostheoarthritis.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation at 3 months | 3 months after surgery
  Experimental tonic pain will be induced by immersing the hand against the side in cold water following the Cold Pressor Test protocol (CPT). CPT will be performed by holding the contralateral hand immersed in water at 12±1 °C up to the wrist for a period of 2 minutes. The evaluation of pain thresholds to pressure will be performed after 45 seconds of immersion at location 1 of the peripatellar region (bilateral) and to the dominant forearm. Both evaluation points have been described in the section on pressure pain thresholds.
  The final value corresponding to the conditioned modulation of pain will be obtained from the difference between the value obtained during the application of the conditioning stimulus and the previous value. The unit of measurement will be in kilopascals (kPa) (conditioned pain modulation = pain threshold at pressure during application of cold - pain threshold at pressure before application of cold).
Conditioned Pain Modulation at 6 months | 6 months after surgery
  Experimental tonic pain will be induced by immersing the hand against the side in cold water following the Cold Pressor Test protocol (CPT). CPT will be performed by holding the contralateral hand immersed in water at 12±1 °C up to the wrist for a period of 2 minutes. The evaluation of pain thresholds to pressure will be performed after 45 seconds of immersion at location 1 of the peripatellar region (bilateral) and to the dominant forearm. Both evaluation points have been described in the section on pressure pain thresholds.
  The final value corresponding to the conditioned modulation of pain will be obtained from the difference between the value obtained during the application of the conditioning stimulus and the previous value. The unit of measurement will be in kilopascals (kPa) (conditioned pain modulation = pain threshold at pressure during application of cold - pain threshold at pressure before application of cold).

SECONDARY OUTCOMES:
Pressure Pain Threshold | 3 and 6 months after surgery
  Eight test sites in the peripatellar region, one control site on tibialis anterior (5 cm distal to the tibial tuberosity) and one control site on the extensor carpi radialis longus (5 cm distal to lateral epicondyle of humerus) were located and marked. The eight sites were located in relation to bone landmark. Site 1: 2 cm distal to the inferior medial edge of patella; site 2: 2 cm distal to the inferior lateral edge of patella; site 3: 3 cm lateral to the mid point on the lateral edge of patella; site 4: 2 cm proximal to the superior lateral edge of patella; site 5: 2 cm proximal to the superior edge of patella; site 6: 2 cm proximal to the superior medial edge of patella; site 7: 3 cm medial to the mid point on the medial edge of patella; site 8: at centre of patella. A hand-held pressure algometer (PAIN TEST™ FPX 50) was used for measuring PPT.
Health Functioning | 3 and 6 months after surgery
  The Spanish version of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used as a measure of health functioning after KA. The WOMAC is a multidimensional scale composed of 24 items grouped into three dimensions: pain (five items), stiffness (two items) and physical function (seventeen items). The WOMAC uses a 5-point Likert scale with responses ranging from 0 - none to 4 - extreme. The final score for the WOMAC was determined by summing the aggregate scores for pain, stiffness, and physical function. The WOMAC is valid and reliable for assessing health functioning in OA participants and is sensitive to changes in health functioning in those who underwent KA.
Pain intensity | 3 and 6 months after surgery
  Pain will be assessed using the reduced version of the McGill Pain Questionnaire (SF-MPQ). The SF*MPQ is a self-administered questionnaire composed of 15 descriptors, 11 of which describe sensory aspects of pain and 4 describe aspects concerning the affective dimension of pain. Each pain descriptor is assessed by scores ranging from 0 to 3 (none, mild, moderate and severe). The pain score is calculated from the sum of the values of the intensity range chosen for each descriptor. The SF-MPQ is considered a valid and reliable assessment tool, routinely used during clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Hospitalari de Vic, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided